CLINICAL TRIAL: NCT01261559
Title: Effect of Displacement During Computed Tomography on Breast Radiation Dose and Image Quality
Brief Title: Breast Displacement and CT Radiation Dose
Acronym: Chrysalis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Claire Kalsch Sandstrom, Fellow, Section of Emergency Radiology, Department of Radiology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 39071
Record Dates: First submitted 2010-12-08; First posted 2010-12-16 (Estimated); Results first posted 2013-11-05 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-06

CONDITIONS: Computed Tomography; Radiation Dosage
Keywords: Computed tomography; Radiation dose; Dose reduction; Breast displacement; Chrysalis device; Image quality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard CT (No Intervention): Women assigned to undergo CT using the standard dose reduction methods (including bismuth shielding and tube current modulation) but without the Chrysalis device.
- Chrysalis CT (Experimental): Women assigned to undergo CT using the standard dose reduction methods (including bismuth shielding and tube current modulation) plus application of the Chrysalis device for breast displacement.
  Interventions: Device: Chrysalis breast displacement device

INTERVENTIONS:
Device: Chrysalis breast displacement device — Chrysalis is a cloth device secured with velcro and buckles around the upper abdomen and chest following manual cephalad breast displacement.
  Arms: Chrysalis CT

SUMMARY:
The primary hypothesis of this study is that breast displacement out of the direct plane of imaging during computed tomography (CT) of the abdomen will reduce effective radiation dose to the female breast. Secondary hypotheses are that image noise and artifacts will also be decreased.

DETAILED DESCRIPTION:
Computed tomography (CT) is a significant source of medical-related radiation, and radiation-related cancer risk is increasingly recognized in the medical and lay community. One of the groups at greatest risk for radiation-induced malignancies is young females due to the radiosensitivity of female breast tissue. Breast tissue frequently lies within the imaging plane for CT of the abdomen with limited gain in diagnostic information. We propose displacing this breast tissue out of the direct imaging plane will decrease unnecessary radiation exposure and may also indirectly improve image quality.

A device called Chrysalis has been designed and received FDA approval for the purposes of displacing female breast tissue during CT.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for CT of the abdomen and pelvis at Harborview Medical Center
* able to provide written informed consent

Exclusion Criteria:

* Inability to provide written consent for self (minor, intubated, sedated, mentally incapacitated, in excessive physical distress)
* Chest or breast surgery within the previous 8 weeks
* Breast implants
* Open wounds to the chest wall
* Fractures of the ribs or spine within the previous 3 months
* Patients requiring oxygen therapy
* Mastectomy
* Breast radiation therapy
* Scarring to the breasts which would prevent displacement
* Claustrophobia is not an absolute exclusion criterion, but patient comfort will be a primary concern.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2010-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire K Sandstrom, MD, Principal Investigator — University of Washington Department of Radiology
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

REFERENCES:
- [Background] Berrington de Gonzalez A, Mahesh M, Kim KP, Bhargavan M, Lewis R, Mettler F, Land C. Projected cancer risks from computed tomographic scans performed in the United States in 2007. Arch Intern Med. 2009 Dec 14;169(22):2071-7. doi: 10.1001/archinternmed.2009.440. PMID 20008689
- [Background] Smith-Bindman R, Lipson J, Marcus R, Kim KP, Mahesh M, Gould R, Berrington de Gonzalez A, Miglioretti DL. Radiation dose associated with common computed tomography examinations and the associated lifetime attributable risk of cancer. Arch Intern Med. 2009 Dec 14;169(22):2078-86. doi: 10.1001/archinternmed.2009.427. PMID 20008690
- [Background] Hurwitz LM, Yoshizumi TT, Reiman RE, Paulson EK, Frush DP, Nguyen GT, Toncheva GI, Goodman PC. Radiation dose to the female breast from 16-MDCT body protocols. AJR Am J Roentgenol. 2006 Jun;186(6):1718-22. doi: 10.2214/AJR.04.1917. PMID 16714665
- [Background] Parker MS, Hui FK, Camacho MA, Chung JK, Broga DW, Sethi NN. Female breast radiation exposure during CT pulmonary angiography. AJR Am J Roentgenol. 2005 Nov;185(5):1228-33. doi: 10.2214/AJR.04.0770. PMID 16247139
- [Background] Pajor L, Kalman E, Koszegi T. Cholesteryl hemisuccinate's inductive effect on membrane rigidization regarding both, its remodelling of the cells' surface receptor pattern and its decreasing the natural killer susceptibility of K-562 cells. Acta Biol Hung. 1991;42(4):371-83. PMID 1841487
- [Background] Yilmaz MH, Albayram S, Yasar D, Ozer H, Adaletli I, Selcuk D, Akman C, Altug A. Female breast radiation exposure during thorax multidetector computed tomography and the effectiveness of bismuth breast shield to reduce breast radiation dose. J Comput Assist Tomogr. 2007 Jan-Feb;31(1):138-42. doi: 10.1097/01.rct.0000235070.50055.e6. PMID 17259846
- [Background] Kang M, Ragan BG, Park JH. Issues in outcomes research: an overview of randomization techniques for clinical trials. J Athl Train. 2008 Apr-Jun;43(2):215-21. doi: 10.4085/1062-6050-43.2.215. PMID 18345348

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment: December 2010 to February 2012, at Harborview Medical Center (inpatient wards, outpatient clinics, and emergency departments)
Pre-assignment Details: All women who were approached for the study were screened for exclusion criteria prior to enrollment.
  110 eligible patients were approached, and 37 declined participation or met exclusion criteria. 1 subject was scanned but TLD readings were clearly erroneous and were therefore excluded. 72 subjects were ultimately included in analyses.
Period: Overall Study
Arm/Group | Standard CT | Chrysalis CT
Started | 36 | 36
Completed | 36 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard CT | Chrysalis CT | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 36 | 72
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (12.9) | 40.3 (12.8) | 40.3 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 36 | 72
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 36 | 36 | 72

OUTCOME MEASURES:

1. Primary Outcome: Skin Entrance Radiation Dose During Computed Tomography (CT)
Description: Skin entrance radiation doses will be measured with Thermoluminescent dosimeters (TLDs) affixed to the subject's chest and breast during CT of the abdomen. TLD #1 is at the inframammary fold, serving as internal control for each subject. Three additional TLDs (#2-4) are affixed to the subject's breast at 3 pre-ascribed locations. The same is done for the right and left breasts (8 TLDs total). TLDs will then be submitted to Landaeur for measurement.
Time Frame: from time potential subject approached about possible enrollment to time device and TLDs were removed, on average 1 hour
Measure: Mean (Standard Deviation); unit: mrad
Arm/Group | Standard CT | Chrysalis CT
Number analyzed (Participants) | 36 | 36
mrad
  Mean entrance skin dose at inframammary fold | 1775 (1634) | 1325 (1158)
  Mean breast entrance skin dose (average TLD2-4) | 625 (677) | 259 (334)

2. Primary Outcome: Relative Skin Entrance Radiation Dose in % During Computed Tomography (CT)
Description: Relative skin entrance dose at the breast (group mean of patient's average skin entrance dose at TLDs 2-4) divided by skin entrance dose at the inframammary TLD (TLD 1) in %. For each patient, doses at TLDs 2-4 were averaged, and then the group mean of this was divided by the group mean at the inframammary TLD, then multiplied by 100 to get % dose. A relative dose of 20% means that the skin entrance dose at the breast was 20% of the skin entrance dose at the inframammary fold.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | Standard CT | Chrysalis CT
Number analyzed (Participants) | 36 | 36
percentage of dose | 37 (30) | 36 (11)
Statistical Analysis 1: Comparison: Standard CT vs Chrysalis CT; Powered to detect difference of 10% at 80% power if 66 or more subjects enrolled; Test type: Superiority or Other; p = 0.003, Regression, Linear; A multivariate linear regression model was fitted for the main outcome of percent relative dose, with age, BMI, and bra cup size as covariates; Mean Difference (Final Values) = 14.2, 95% CI 2-sided [4 to 25], Standard Deviation 10

3. Secondary Outcome: CT Image Noise
Description: To evaluate image noise, mean of the Standard deviation (SD) of the pixel values, measured in Hounsfield units (HU), will be measured in Picture Archiving and Communication System (PACS) using a region of interest (ROI) measuring 90-110 mm^2 in size drawn over each of these body regions: hepatic dome, spleen, renal cortex, retroperitoneal fat, subcutaneous fat, paraspinal muscles, and if present, breast tissue, avoiding vascular structures in each case. SD for ROI measuring 90-110 mm^2 in size will also be drawn over the aorta and inferior vena cava (IVC), remote from contrast mixing artifact, and over medullary bone of the spine.
  HU is the linear scale by which digital image data are displayed in PACS and reflect relative attenuation compared to distilled water at a standard temperature and pressure (STP) (defined as 0 HU) and of pure air at STP (defined as -1000HU). Within a drawn ROI, the PACS will give the mean attenuation (in HU) and the standard deviation of HU (reflecting
Time Frame: two months
Population: In some cases, a reliable measurement of noise could not be measured on the location. For example, if the breast was not included on the CT, breast noise could not be measured (12 controls and 21 Chrysalis). Too little retroperitoneal or subcutaneous fat was present to draw the relevant ROI in 1 control and 1 Chrysalis subject, respectively.
Measure: Mean (Standard Deviation); unit: Hounsfield units
Arm/Group | Standard CT | Chrysalis CT
Number analyzed (Participants) | 36 | 36
Hounsfield units
  Liver dome | 17.1 (5.9) | 16.4 (6.9)
  Spleen: number analyzed (Participants) | 36 | 35
  Spleen | 23.2 (8.1) | 21.1 (7.3)
  Kidney | 26.8 (8.0) | 24.5 (6.8)
  Aorta (without mixing artifact) | 19.7 (5.0) | 21.1 (7.26)
  IVC (without mixing artifact): number analyzed (Participants) | 36 | 34
  IVC (without mixing artifact) | 21.1 (5.1) | 22.9 (5.7)
  Retroperitoneal fat: number analyzed (Participants) | 35 | 36
  Retroperitoneal fat | 24.4 (7.9) | 23.4 (7.0)
  Subcutaneous fat: number analyzed (Participants) | 36 | 35
  Subcutaneous fat | 13.3 (4.0) | 12.9 (3.5)
  Medullary Bone of Spine | 31.2 (7.4) | 34.8 (18.2)
  Paraspinal muscle | 19.8 (7.7) | 17.9 (5.6)
  Breast (if imaged): number analyzed (Participants) | 24 | 15
  Breast (if imaged) | 26.0 (9.9) | 26.1 (11.1)

4. Secondary Outcome: Number of Participants With Presence of Artifacts Based on CT Image Quality
Description: CT images acquired will be reviewed for the presence of artifacts that might be attributed to the displacement device or to the presence of the breast tissue.
  To evaluate for artifacts, the exam will be qualitatively reviewed by a board certified radiologist for imaging artifacts, such as streak artifact. It will be noted on a per participant basis whether any imaging artifacts are identified.
Time Frame: two months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard CT | Chrysalis CT
Number analyzed (Participants) | 36 | 36
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: from time potential subject was approached about possible enrollment to the time when the device and TLDs were removed.
Arm/Group | Standard CT | Chrysalis CT
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No